CLINICAL TRIAL: NCT03238001
Title: Evaluation of DCTclock™ as a Cognitive Assessment Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Digital Cognition Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DCT032
Record Dates: First submitted 2017-07-27; First posted 2017-08-03 (Actual); Results first posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Cognitive Function
Keywords: Cognitive assessment; Cognition; Clock Test

STUDY DESIGN:
Intervention Model Description: This study uses a paired design in which each subject undergoes blinded testing by separate testers administering DCTclock and a battery of reference standard tests to determine cognitive state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All qualified participants (Experimental): Participants received DCTclock, Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), and a battery of other traditional pen and paper neuropsychological assessments.
  Interventions: Device: DCTclock

INTERVENTIONS:
Device: DCTclock — DCTclock is a quick and non-invasive test that measures cognitive function based on a computerized algorithmic analysis of the entire drawing process and output of a well-established cognitive assessment called The Clock Drawing Test (CDT).

SUMMARY:
The overall objective of this study is to demonstrate the safety and effectiveness of DCTclock as an adjunctive tool for use by clinicians to evaluate cognitive function in adults aged 55-95.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 55 to 95 years old.

Exclusion Criteria:

* Ineligible for written informed consent.
* Physical impairment of the writing hand.
* Impaired manual dexterity.
* Impaired vision.
* Under the influence of recreational drugs or alcohol at the time of the visit.
* Current or recent participation in a clinical trial that includes the use of a drug or intervention to alter cognitive function.
* Recent cognitive testing.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonia H Holway, Ph.D., Study Director — Digital Cognition Technologies, Inc.
Locations (1):
- Compass Research, Maitland, Florida, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD

REFERENCES:
- [Background] Lamar M, Ajilore O, Leow A, Charlton R, Cohen J, GadElkarim J, Yang S, Zhang A, Davis R, Penney D, Libon DJ, Kumar A. Cognitive and connectome properties detectable through individual differences in graphomotor organization. Neuropsychologia. 2016 May;85:301-9. doi: 10.1016/j.neuropsychologia.2016.03.034. Epub 2016 Mar 30. PMID 27037044
- [Background] Souillard-Mandar W, Davis R, Rudin C, Au R, Libon DJ, Swenson R, Price CC, Lamar M, Penney DL. Learning Classification Models of Cognitive Conditions from Subtle Behaviors in the Digital Clock Drawing Test. Mach Learn. 2016 Mar;102(3):393-441. doi: 10.1007/s10994-015-5529-5. Epub 2015 Oct 20. PMID 27057085
- [Background] Cohen J, Penney DL, Davis R, Libon DJ, Swenson RA, Ajilore O, Kumar A, Lamar M. Digital Clock Drawing: differentiating "thinking" versus "doing" in younger and older adults with depression. J Int Neuropsychol Soc. 2014 Oct;20(9):920-8. doi: 10.1017/S1355617714000757. Epub 2014 Sep 15. PMID 25222513
- [Background] Davis R, Libon DJ, Au R, Pitman D, Penney DL. THink: Inferring Cognitive Status from Subtle Behaviors. Proc AAAI Conf Artif Intell. 2014 Jul;2014:2898-2905. PMID 27066307

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at one site in the US.
Pre-assignment Details: 450 participants were enrolled. 14 did not meet screening criteria.
Groups:
- All Qualified Participants: Participants received the DCTclock test and a battery of other traditional, pen and paper, neuropsychological assessments.
Period: Visit 1 (Primary Endpoint Cohort)
Arm/Group | All Qualified Participants
Started | 436
Completed | 432
Not Completed | 4
Not completed — Protocol Violation | 2
Not completed — Unanalyzable test result | 2
Period: Visit 2 (Secondary Endpoint Cohort)
Arm/Group | All Qualified Participants
Started | 432
Completed | 403
Not Completed | 29
Not completed — Lost to Follow-up | 16
Not completed — Unanalyzable test result | 2
Not completed — Withdrawal by Subject | 3
Not completed — Met exclusion criteria at visit 2 | 3
Not completed — Study completion | 1
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants enrolled in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.94 (8.78)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 114
  Female | 333
  Unknown or Other | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38
  Not Hispanic or Latino | 405
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 105
  White | 329
  More than one race | 4
  Unknown or Not Reported | 6
Handedness [Count of Participants; unit: Participants]
  Right handed | 396
  Left handed | 34
  Ambidextrous | 13
  Other or unknown | 7
Highest education level attained [Count of Participants; unit: Participants]
  College Degree + | 148
  High School and some college | 141
  High school | 106
  Less than high school | 45
  Unknown | 10

OUTCOME MEASURES:

1. Primary Outcome: Non-Inferiority of DCTclock Compared to Mini-Mental State Examination (MMSE)
Description: The primary analysis will assess agreement between DCTclock and the Montreal Cognitive Assessment (MoCA) and compare it to the agreement between the MMSE and MoCA at visit 1.
Time Frame: Visit 1 (day 1)
Population: The Evaluable Population includes all qualified participants undergoing cognitive testing with DCTclock, MMSE, and MoCA who completed visit 1.
Measure: Number (90% Confidence Interval); unit: Difference in Quadratic Weighted Kappas
Groups:
- Primary Endpoint (Evaluable) Population: Participants received DCTclock, MMSE, MoCA, and a battery of other traditional pen and paper neuropsychological assessments.
Arm/Group | Primary Endpoint (Evaluable) Population
Number analyzed (Participants) | 432
Difference in Quadratic Weighted Kappas | -0.035 [-0.12 to 0.05]
Statistical Analysis 1: Comparison: Primary Endpoint (Evaluable) Population; A two-one-sided tests approach was taken, where, prior to analysis, it was determined that a delta (equivalence margin) of 0.20 would be considered a significant difference between the DCTclock/MoCA kappa and the MMSE/MoCA kappa. The reasoning behind this determination can be found in the study's statistical analysis plan; Test type: Non-Inferiority — In order to show non-inferiority, a lower 90% confidence limit (CL) for the difference in kappa scores would need to be greater than or equal to -0.20. The 90% confidence interval was calculated based on 5000 bootstrapped differences in kappa scores; Lower 90% CL for difference in Kappas = -0.12, 90% CI 2-sided [-0.12 to 0.05] — 90% CI for Kappa of DCTclock/MoCA - Kappa of MMSE/MoCA (estimated with bootstrap method using 5000 bootstraps)

2. Secondary Outcome: Quadratic Weighted Kappa on Primary Endpoints
Description: Quadratic weighted Cohen's kappa with 95% CI between DCTclock and MoCA, as well as between MMSE and MoCA.
Time Frame: Visit 1 (day 1)
Measure: Number (95% Confidence Interval); unit: Quadratic Weighted Kappa
Groups:
- DCTclock: Participants received DCTclock and MoCA on their first visit.
- MMSE: Participants received MMSE and MoCA on their first visit.
Arm/Group | DCTclock | MMSE
Number analyzed (Participants) | 432 | 432
Quadratic Weighted Kappa | 0.40 [0.32 to 0.49] | 0.44 [0.36 to 0.52]

3. Secondary Outcome: Percent Agreement on Primary Endpoints
Description: Positive percent agreement, version A (treating the "Indeterminate" group as "Unimpaired") and version B (removing the "Indeterminate" group from the analysis), and negative percent agreement version A and version B. These were calculated for the DCTclock/MoCA classification table as well as the MMSE/MoCA classification table. 95% CI were also calculated and compared between the two classification tables' calculations.
Time Frame: Visit 1 (day 1)
Population: Version A treats the "Indeterminate" group as "Unimpaired", while version B removes the "Indeterminate" group from the analysis. Thus, the analysis population for version B is smaller than the overall analysis population.
Measure: Number (95% Confidence Interval); unit: Percent Agreement
Arm/Group | DCTclock | MMSE
Number analyzed (Participants) | 432 | 432
Percent Agreement
  Positive - Version A | 0.64 [0.57 to 0.71] | 0.56 [0.49 to 0.63]
  Positive - Version B: number analyzed (Participants) | 268 | 273
  Positive - Version B | 0.78 [0.71 to 0.84] | 0.69 [0.62 to 0.76]
  Negative - Version A | 0.74 [0.69 to 0.80] | 0.83 [0.78 to 0.87]
  Negative - Version B: number analyzed (Participants) | 268 | 273
  Negative - Version B | 0.73 [0.64 to 0.81] | 0.88 [0.81 to 0.93]

4. Secondary Outcome: Regression Coefficients on Primary Endpoints
Description: Linear and rank-linear regression coefficients (slope, intercept) and 95% CI for DCTclock regressed on MoCA as well as for the MMSE regressed on MoCA.
Time Frame: Visit 1 (day 1)
Measure: Number (95% Confidence Interval); unit: Regression Coefficients
Arm/Group | DCTclock | MMSE
Number analyzed (Participants) | 432 | 432
Regression Coefficients
  Linear - Intercept | 19.35 [18.64 to 20.07] | -5.03 [-8.73 to -1.32]
  Linear - Slope | 0.07 [0.06 to 0.08] | 1.03 [0.90 to 1.17]
  Rank-Linear - Intercept | 107.75 [87.37 to 128.12] | 96.45 [76.43 to 116.48]
  Rank-Linear - Slope | 0.50 [0.42 to 0.58] | 0.55 [0.47 to 0.63]

5. Secondary Outcome: Correlation Coefficients on Primary Endpoints
Description: Pearson and Spearman correlation coefficients between DCTclock and MoCA as well as between MMSE and MoCA.
Time Frame: Visit 1 (day 1)
Measure: Number (95% Confidence Interval); unit: Correlation Coefficients
Arm/Group | DCTclock | MMSE
Number analyzed (Participants) | 432 | 432
Correlation Coefficients
  Pearson | 0.53 [0.46 to 0.60] | 0.59 [0.53 to 0.65]
  Spearman | 0.50 [0.43 to 0.57] | 0.55 [0.48 to 0.61]

6. Secondary Outcome: Quadratic Weighted Kappa on Secondary Endpoints (Test-Retest Reliability)
Description: Quadratic weighted Cohen's Kappa statistics were calculated for both DCTclock and MMSE test-retest data (visit 1 vs visit 2).
Time Frame: Visit 1 and visit 2, occurring 1-4 weeks apart
Measure: Number (95% Confidence Interval); unit: Quadratic Weighted Cohen's Kappa
Groups:
- DCTclock: Participants received DCTclock on their first and second visits, occurring 1-4 weeks apart.
- MMSE: Participants received MMSE on their first and second visits, occurring 1-4 weeks apart.
Arm/Group | DCTclock | MMSE
Number analyzed (Participants) | 403 | 403
Quadratic Weighted Cohen's Kappa | 0.53 [0.45 to 0.60] | 0.48 [0.39 to 0.56]

7. Secondary Outcome: Percent Agreement on Secondary Endpoints (Test-retest Reliability)
Description: Positive percent agreement version A (treating the "Indeterminate" group as "Unimpaired") and version B (removing the "Indeterminate" group from the analysis), negative percent agreement version A and version B, indeterminate percent agreement, and unimpaired percent agreement.
Time Frame: Visit 1 and visit 2, occurring 1-4 weeks apart
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percent Agreement
Arm/Group | DCTclock | MMSE
Number analyzed (Participants) | 403 | 403
Percent Agreement
  Positive - Version A | 0.73 [0.66 to 0.80] | 0.74 [0.65 to 0.82]
  Positive - Version B: number analyzed (Participants) | 257 | 283
  Positive - Version B | 0.85 [0.77 to 0.90] | 0.84 [0.75 to 0.90]
  Negative - Version A | 0.76 [0.70 to 0.81] | 0.80 [0.75 to 0.84]
  Negative - Version B: number analyzed (Participants) | 257 | 283
  Negative - Version B | 0.81 [0.74 to 0.87] | 0.78 [0.72 to 0.84]
  Indeterminate | 0.21 [0.14 to 0.31] | 0.27 [0.17 to 0.39]
  Unimpaired | 0.61 [0.54 to 0.68] | 0.63 [0.57 to 0.69]

8. Secondary Outcome: Regression Coefficients on Secondary Endpoints (Test-retest Reliability)
Description: Deming, linear, and rank-linear correlation coefficients (intercept, slope) were calculated for visit 1 regressed on visit 2 for both DCTclock and MMSE.
Time Frame: Visit 1 and visit 2, occurring 1-4 weeks apart
Measure: Number (95% Confidence Interval); unit: Regression Coefficients
Arm/Group | DCTclock | MMSE
Number analyzed (Participants) | 403 | 403
Regression Coefficients
  Deming - Intercept | 8.77 [3.07 to 14.46] | 2.96 [-0.46 to 6.37]
  Deming - Slope | 0.93 [0.85 to 1.00] | 0.91 [0.79 to 1.03]
  Linear - Intercept | 25.03 [20.58 to 29.48] | 10.88 [8.96 to 12.80]
  Linear - Slope | 0.66 [0.60 to 0.73] | 0.62 [0.55 to 0.69]
  Rank-Linear - Intercept | 66.48 [49.51 to 83.46] | 91.16 [72.43 to 109.89]
  Rank-Linear - Slope | 0.67 [0.60 to 0.74] | 0.55 [0.47 to 0.63]

9. Secondary Outcome: Correlation Coefficients on Secondary Endpoints (Test-retest Reliability)
Description: Pearson and Spearman correlation coefficients were calculated between visit 1 and visit 2 for DCTclock and MMSE, along with 95% CI.
Time Frame: Visit 1 and visit 2, occurring 1-4 weeks apart
Measure: Number (95% Confidence Interval); unit: Correlation Coefficients
Arm/Group | DCTclock | MMSE
Number analyzed (Participants) | 403 | 403
Correlation Coefficients
  Pearson | 0.70 [0.64 to 0.75] | 0.67 [0.61 to 0.72]
  Spearman | 0.67 [0.60 to 0.73] | 0.56 [0.47 to 0.62]

10. Other Pre Specified Outcome: Construct Validity of DCTclock as Measured by the Comparison of DCTclock Results to the Results of a Battery of Neuropsychological Assessments
Description: The goal of this analysis is to assess the construct validity of DCTclock. Specifically, the goal is to compare scores from the administration of DCTclock to the visit 1 administration of a battery of neuropsychological tests, to characterize the psychometric properties of DCTclock, and to compare those properties to the properties of MMSE.
Time Frame: Visit 1 (day 1)
Population: Includes all qualified participants who completed testing at visit 1 and had evaluable data for each test analyzed. Roughly half of the population was administered the full neuropsychological battery. The remainder completed a partial battery (see protocol for details).
Measure: Number (95% Confidence Interval); unit: Correlation Coefficient
Groups:
- DCTclock; MMSE: Participants received DCTclock, MMSE, MoCA, and a battery of other traditional pen and paper neuropsychological assessments.
Arm/Group | DCTclock | MMSE
Number analyzed (Participants) | 432 | 432
Correlation Coefficient
  MMSE | 0.50 [0.42 to 0.57] | NA [NA to NA] — Row = Column (correlation of MMSE to MMSE)
  MoCA | 0.53 [0.46 to 0.60] | 0.59 [0.53 to 0.65]
  Benton Judgment of Line Orientation: number analyzed (Participants) | 194 | 194
  Benton Judgment of Line Orientation | 0.34 [0.21 to 0.46] | 0.36 [0.23 to 0.48]
  Delis-Kaplan Executive Function- Letter Fluency: number analyzed (Participants) | 195 | 195
  Delis-Kaplan Executive Function- Letter Fluency | 0.36 [0.23 to 0.48] | 0.34 [0.21 to 0.46]
  Delis-Kaplan Executive Function-Category Fluency: number analyzed (Participants) | 194 | 194
  Delis-Kaplan Executive Function-Category Fluency | 0.39 [0.27 to 0.50] | 0.37 [0.24 to 0.49]
  Delis-Kaplan Executive Function-Category Switching: number analyzed (Participants) | 194 | 194
  Delis-Kaplan Executive Function-Category Switching | 0.30 [0.16 to 0.42] | 0.38 [0.25 to 0.49]
  Delis-Kaplan Executive Function- Switch Accuracy: number analyzed (Participants) | 194 | 194
  Delis-Kaplan Executive Function- Switch Accuracy | 0.26 [0.13 to 0.39] | 0.36 [0.24 to 0.48]
  Rey-Osterrieth Complex Figure- Copy: number analyzed (Participants) | 182 | 182
  Rey-Osterrieth Complex Figure- Copy | 0.44 [0.31 to 0.55] | 0.43 [0.31 to 0.55]
  Rey-Osterrieth Complex Figure- Immediate: number analyzed (Participants) | 194 | 194
  Rey-Osterrieth Complex Figure- Immediate | 0.43 [0.31 to 0.54] | 0.31 [0.17 to 0.43]
  Rey-Osterrieth Complex Figure- Delayed: number analyzed (Participants) | 193 | 193
  Rey-Osterrieth Complex Figure- Delayed | 0.39 [0.26 to 0.50] | 0.28 [0.14 to 0.40]
  Rey-Osterrieth Complex Figure- Immediate Retention: number analyzed (Participants) | 193 | 193
  Rey-Osterrieth Complex Figure- Immediate Retention | 0.22 [0.08 to 0.35] | 0.08 [-0.06 to 0.22]
  Rey-Osterrieth Complex Figure- Delayed Retention: number analyzed (Participants) | 190 | 190
  Rey-Osterrieth Complex Figure- Delayed Retention | -0.06 [-0.20 to 0.09] | 0.03 [-0.11 to 0.17]
  Rey-Osterrieth Complex Figure- Organization: number analyzed (Participants) | 193 | 193
  Rey-Osterrieth Complex Figure- Organization | 0.29 [0.16 to 0.42] | 0.25 [0.11 to 0.38]
  WAIS-IV Digit Span: number analyzed (Participants) | 431 | 431
  WAIS-IV Digit Span | 0.32 [0.23 to 0.40] | 0.48 [0.40 to 0.55]
  WAIS-IV Block Design: number analyzed (Participants) | 190 | 190
  WAIS-IV Block Design | 0.39 [0.27 to 0.51] | 0.42 [0.29 to 0.53]
  Trail Making Part A: number analyzed (Participants) | 431 | 431
  Trail Making Part A | 0.48 [0.40 to 0.55] | 0.45 [0.38 to 0.53]
  Trail Making Part B: number analyzed (Participants) | 420 | 420
  Trail Making Part B | 0.49 [0.41 to 0.56] | 0.51 [0.44 to 0.58]
  Geriatric Depression Scale: number analyzed (Participants) | 194 | 194
  Geriatric Depression Scale | -0.11 [-0.24 to 0.03] | -0.04 [-0.18 to 0.10]
  Symbol Digit Modalities: number analyzed (Participants) | 195 | 195
  Symbol Digit Modalities | 0.51 [0.39 to 0.60] | 0.49 [0.37 to 0.59]
  Hamilton-Veale Contrast Sensitivity - Left | 0.12 [0.03 to 0.22] | 0.10 [0.01 to 0.19]
  Hamilton-Veale Contrast Sensitivity- Right | 0.09 [-0.00 to 0.18] | 0.17 [0.08 to 0.26]
  Hamilton-Veale Contrast Sensitivity- Binocular | 0.24 [0.14 to 0.32] | 0.21 [0.11 to 0.29]
  Purdue Peg Board- Left hand | 0.32 [0.24 to 0.41] | 0.16 [0.07 to 0.25]
  Purdue Peg Board- Right hand | 0.35 [0.27 to 0.43] | 0.22 [0.12 to 0.30]
  Purdue Peg Board- Bimanual | 0.36 [0.28 to 0.44] | 0.25 [0.16 to 0.34]

11. Other Pre Specified Outcome: Incidence of Serious Device-related Adverse Events [Safety]
Description: Incidence of serious device-related adverse events.
Time Frame: Visit 1 and visit 2, occuring 1-4 weeks apart
Population: All qualified participants who completed at least one DCTclock test.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Participants received DCTclock, MMSE, MoCA, and a battery of other traditional pen and paper neuropsychological assessments.
Arm/Group | All Participants
Number analyzed (Participants) | 432
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at each study visit. The second (final) study visit occurred one to four weeks after the first visit, therefore, adverse event data was collected for a period of one to four weeks.
Groups:
- All Participants: Participants received DCTclock, MMSE, MoCA, and a battery of other traditional, pen and paper neuropsychological assessments.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/436
Serious Adverse Events (participants affected / at risk) | 1/436
Other Adverse Events (participants affected / at risk) | 0/436
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=436)
Bone fracture (Injury, poisoning and procedural complications) | 1 (1) — Accidental fall resulting in bone fracture.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT03238001/SAP_000.pdf
  • Study Protocol (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT03238001/Prot_001.pdf